CLINICAL TRIAL: NCT02015351
Title: Intravitreal Bevacizumab for the Treatment of Choroidal Neovascularization in Vogt-Koyanagi-Harada Disease - A Prospective Study
Brief Title: Intravitreal Bevacizumab for the Treatment of CNV in VKH Disease - A Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Joyce Hisae Yamamoto, MD, PhD, Coordinator of the Uveitis Service, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brazilian VKH Study Group
Record Dates: First submitted 2013-12-05; First posted 2013-12-19 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Choroidal Neovascularization
Keywords: Choroidal neovascularization; Vogt Koyanagi Harada Disease; Inflammatory choroidal neovascularization; Anti-VEGF
MeSH Terms: conditions — Choroidal Neovascularization; Uveomeningoencephalitic Syndrome | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-VEGF and Immunosuppression (Experimental): Bevacizumab: Dosage 1.25mg/0.05ml; Frequency monthly injections; Duration at least 3 months.
  Immunosuppression: cyclosporine and/or azathioprine
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — Injection technique: After lid speculum insertion and irrigation of the conjunctiva with 5% povidone-iodine, 0,05ml of bevacizumab will be inserted through the pars plana 3.5mm to 4.0mm posterior to the surgical limbus using a 30 gauge needle. After injection, topical antibiotics will be immediately applied in the injected eye. Immunosuppression: Corticosteroids will be prescribed (1mg/Kg/d) with tapering along 5 months. Immunosuppressive drug of choice is cyclosporine (3-5mg/Kg/d). In case of contraindication to cyclosporine use, azathioprine or mycophenolate mofetil will be prescribed.
  Other Names: Bevacizumab (Avastin;Genentech Inc,USA)

SUMMARY:
Efficacy of monthly intravitreal anti-vascular endothelial growth factor (VEGF) associated to systemic immunosuppression in patients with Vogt-Koyanagi-Harada Disease and choroidal neovascularization. Minimum follow-up 12 months. Endpoints: 6 and 12 months of follow-up. Outcome measures: improvement of VA, decrease in central foveal thickness as measured by Optical Coherence Tomography (OCT) and absence of intra/subretinal fluid.

DETAILED DESCRIPTION:
Choroidal neovascularization (CNV) in Vogt-Koyanagi-Harada (VKH) disease is associated with poor visual prognosis. Several treatments have been suggested, though there is still no standard therapy. CNV diagnosis will be based on fundus biomicroscopy (presence of serous retinal detachment with or without retinal hemorrhages), fluorescein angiography (FA) (presence of early phase hyperfluorescence with late phase leakage) and OCT findings (hyperreflective lesion related to a CNV complex with serous foveal detachment or intraretinal fluid with increased foveal thickness). Inflammation will be considered active if anterior chamber cells or optic disc leakage in FA is observed. Each patient will undergo a complete clinical exam, including best corrected visual acuity (VA) (Snellen charts). Once active CNV is identified, a loading dose of 3 injections of IV bevacizumab will be proceeded monthly and systemic immunosuppression will be introduced or intensified. After the first 3 injections, the patient will be clinically examined and OCT will be proceeded monthly. The persistence of intra/subretinal fluid in the OCT will indicate one more IV bevacizumab injection. Immunosuppression status evaluation will be done at 3, 6, 9 and 12 months of follow up and intensification will be done if inflammatory signs or persistence of intraretinal fluid is observed. Presence of intra/subretinal fluid and manual measurement of retina central foveal thickness (CFT) will be proceeded in horizontal scan by the same examiner.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Vogt-Koyanagi-Harada disease based on Revised Diagnostic Criteria presented by the International Committee on VKH disease in 2001;
2. Presence of choroidal neovascularization identified by fundus biomicroscopy, fluorescein angiography and OCT.

Exclusion Criteria:

* Media opacities precluding posterior segment exam, ametropia over 5 dioptries, glaucoma (defined as a disease with characteristic damage at the optic nerve or characteristic visual field defect with compatible nerve fiber layer lesion), Age related Macular degeneration, impossibility to increase immunosuppression.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Visual Acuity change | 6 months
  Visual Acuity will be measured using Snellen charts with best refraction by the same examiner.
Change in central foveal thickness | 6 months
  Central foveal thickness will be measured manually using the caliper by the same examiner. Measurements will be proceeded from the Bruch's membrane till the internal limiting membrane and comparison with previous measurement will be done.
Presence or absence of intra/subretinal fluid in OCT | 6 months
  OCT will be analyzed at 6 and 12 months for the presence of intra or subretinal fluid.

SECONDARY OUTCOMES:
Visual Acuity change | 12 months
  Visual Acuity will be measured using Snellen charts with best refraction by the same examiner.
Change in Central Foveal Thickness | 12 months
  Central foveal thickness will be measured manually using the caliper by the same examiner. Measurements will be proceeded from the Bruch's membrane till the internal limiting membrane and comparison with previous measurement will be done.
Presence or Absence of Intra/Subretinal fluid in OCT | 12 months
  OCT will be analyzed at 6 and 12 months for the presence of intra or subretinal fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce H Yamamoto, MD, Principal Investigator — University of Sao Paulo School of Medicine Ophthalmology; Viviane M Sakata, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas- University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Perentes Y, Van Tran T, Sickenberg M, Herbort CP. Subretinal neovascular membranes complicating uveitis: frequency, treatments, and visual outcome. Ocul Immunol Inflamm. 2005 Apr-Jun;13(2-3):219-24. doi: 10.1080/09273940490518883. PMID 16019682
- [Result] Rouvas A, Petrou P, Douvali M, Ntouraki A, Vergados I, Georgalas I, Markomichelakis N. Intravitreal ranibizumab for the treatment of inflammatory choroidal neovascularization. Retina. 2011 May;31(5):871-9. doi: 10.1097/IAE.0b013e3182003ca8. PMID 21358461
- [Result] Adan A, Mateo C, Navarro R, Bitrian E, Casaroli-Marano RP. Intravitreal bevacizumab (avastin) injection as primary treatment of inflammatory choroidal neovascularization. Retina. 2007 Nov-Dec;27(9):1180-6. doi: 10.1097/IAE.0b013e31815e9834. PMID 18046222
- [Result] Wu L, Evans T, Saravia M, Schlaen A, Couto C. Intravitreal bevacizumab for choroidal neovascularization secondary to Vogt-Koyanagi-Harada syndrome. Jpn J Ophthalmol. 2009 Jan;53(1):57-60. doi: 10.1007/s10384-008-0600-4. Epub 2009 Jan 30. PMID 19184312
- [Result] Kolomeyer AM, Roy MS, Chu DS. The use of intravitreal ranibizumab for choroidal neovascularization associated with vogt-koyanagi-harada syndrome. Case Rep Med. 2011;2011:747648. doi: 10.1155/2011/747648. Epub 2011 Aug 3. PMID 21826150
- [Result] Tran TH, Fardeau C, Terrada C, Ducos De Lahitte G, Bodaghi B, Lehoang P. Intravitreal bevacizumab for refractory choroidal neovascularization (CNV) secondary to uveitis. Graefes Arch Clin Exp Ophthalmol. 2008 Dec;246(12):1685-92. doi: 10.1007/s00417-008-0906-4. Epub 2008 Aug 6. PMID 18682970
- [Result] Nowilaty SR, Bouhaimed M; Photodynamic Therapy Study Group. Photodynamic therapy for subfoveal choroidal neovascularisation in Vogt-Koyanagi-Harada disease. Br J Ophthalmol. 2006 Aug;90(8):982-6. doi: 10.1136/bjo.2006.091538. Epub 2006 May 10. PMID 16687455
- [Result] Mansour AM, Arevalo JF, Ziemssen F, Mehio-Sibai A, Mackensen F, Adan A, Chan WM, Ness T, Banker AS, Dodwell D, Chau Tran TH, Fardeau C, Lehoang P, Mahendradas P, Berrocal M, Tabbarah Z, Hrisomalos N, Hrisomalos F, Al-Salem K, Guthoff R. Long-term visual outcomes of intravitreal bevacizumab in inflammatory ocular neovascularization. Am J Ophthalmol. 2009 Aug;148(2):310-316.e2. doi: 10.1016/j.ajo.2009.03.023. Epub 2009 May 9. PMID 19427992